CLINICAL TRIAL: NCT03172325
Title: A Phase III, Randomized, Two-armed, Double-blind, Parallel, Active Controlled Clinical Trial to Determine the Non-inferior Efficacy and Safety of CinnoRA® (Adalimumab, CinnaGen Co.) Versus Humira® for Treatment of Active RA
Brief Title: Study to Demonstrate Non-Inferior Efficacy and Safety of CinnoRA® Versus Humira® for Treatment of Active RA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADA.CIN.AJ94; IRCT2015030321315N1 (Other: Food And Drug Administration of The Islamic Republic of Iran)
Record Dates: First submitted 2017-05-24; First posted 2017-06-01 (Actual); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Active Rheumatoid Arthritis
MeSH Terms: interventions — Adalimumab; Methotrexate; Folic Acid; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CinnaGen adalimumab (Experimental): CinnoRA® (adalimumab Prefilled Syringe produced by CinnaGen Company) 40 mg/0.8 ml Every other week 40 mg Adalimumab, will be subcutaneously administered to rheumatic patients during six months. Along with, 15 mg weekly methotrexate, at least 1 mg daily Folic acid and 7.5 mg daily Prednisolone over six months.
  Interventions: Drug: Adalimumab; Drug: Methotrexate; Drug: Folic Acid; Drug: Prednisolone
- AbbVie adalimumab (Active Comparator): Humira® (adalimumab Prefilled Syringe produced by AbbVie Company) 40 mg/0.8 ml Every other week 40 mg Adalimumab, will be subcutaneously administered to rheumatic patients during six months. Along with, 15 mg weekly methotrexate, at least 1 mg daily Folic acid and 7.5 mg daily Prednisolone over six months.
  Interventions: Drug: Adalimumab; Drug: Methotrexate; Drug: Folic Acid; Drug: Prednisolone

INTERVENTIONS:
Drug: Adalimumab — 40 mg Adalimumab every other week is administered subcutaneously to all the patients.
Drug: Methotrexate — 15 mg Methotrexate is weekly administered to all the patients.
Drug: Folic Acid — At least 1 mg Folic acid is daily administered to all the patients.
Drug: Prednisolone — 7.5 mg Prednisolone is daily administered to all the patients.

SUMMARY:
The purpose of this study is to compare the efficacy and safety of adalimumab produced by CinnaGen company and AbbVie adalimumab in subjects with active Rheumatoid Arthritis. Patients with the diagnosis of active Rheumatoid arthritis according to EULAR criteria (European League Against Rheumatism) aged between 18 to 75 years will be included. This study is a Phase III, randomized, two arms, double-blind (patient and assessor blinded), parallel active-controlled non-inferiority clinical trial. The eligible patients are randomized in a 1:1 ratio to receive CinnoRA® or Humira®. Every two weeks, 40 mg of either of the drugs will be administered to each patient subcutaneously along with methotrexate (15 mg/week), folic acid (1 mg/day), and prednisolone (7.5 mg/day) over six months.

The primary objective of the study is to compare the efficacy of test- adalimumab (CinnoRA®) and the reference adalimumab (Humira®) in patients with moderately to severely active rheumatoid arthritis regarding the evaluation of EULAR criteria based on Disease activity score (DAS).

The secondary objectives of this study are:

* To further compare the efficacy of test- adalimumab to reference adalimumab
* To assess the safety of test- adalimumab compared to reference adalimumab

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy and safety of Adalimumab produced by CinnaGen company and AbbVie adalimumab in subjects with active rheumatoid arthritis. Patients with the diagnosis of active rheumatoid arthritis according to EULAR criteria (European League Against Rheumatism) aged between 18 to 75 years will be included. This study is a Phase III, randomized, two arms, double-blind (patient and assessor blinded), parallel active-controlled non-inferiority clinical trial. The eligible patients will be randomized in a 1:1 ratio to receive CinnoRA® or Humira®. Every two weeks, 40 mg of either of the drugs will be administered to each patient subcutaneously along with methotrexate (15 mg/week), folic acid (1 mg/day), and prednisolone (7.5 mg/day) over six months.

Physical examinations, vital signs, disease activity, and laboratory parameters will be evaluated for patients at baseline and 3 and 6-month visits. The incidence of adverse events at each visit will be recorded based on patients' reports, vital signs, physical examinations, and laboratory tests.

The trial is reviewed by food and drug administration of Iran. The protocol, case report form (CRF), information for patients, and informed consent form are submitted to the ethics committees responsible for review and approval purposes, according to national regulatory guidelines.

In this study, no patient will be recruited without an informed consent form. All the informed consent forms which will be signed by the patients will have two copies so that patients can receive a copy of it.

Determination of sample size:

The outcome measures of this study are changes in composite scores defined by the European League against Rheumatism (EULAR) and the American College of Rheumatology criterions. The CinnoRA® group proportion is assumed to be 0.7100 under the null hypothesis of inferiority. If the response rate of CinnoRA® is at most 18% worse than Humira® (δ = -0.18) (non-inferiority margin), it will be considered to be non-inferior. Sample size 64 in both Humira and CinnoRA® groups yields 90% power to detect non-inferiority margin. The significance level of the test is targeted at 0.0250 (The significance level actually achieved by this design is 0.0284).

DATA QUALITY ASSURANCE:

CinnaGen Company conducts clinical trials according to procedures that incorporate the ethical principles of good clinical practice (GCP). Accurate and reliable data collection is assured by verification and cross-check of the CRFs against the patient's records by clinical monitors, and the maintenance of a drug-dispensing log by the center.

Principle and coordinating investigators, contract research organization (CRO) coordinators and sponsor personnel attend the investigator meetings, and at the end, they receive a GCP certificate.

CRO coordinators and one sponsor attend the Site Initiation Visit (SIV) meetings. Protocol and GCP principles are reviewed by coordinating investigator of each site, and also the needed information for completing CRF and Trial Master File (TMF) forms are explained.

Monitoring by CRO will be performed in 30% and 70% of study progress and at the end of the study. In the monitoring sessions, some sponsor personnel will audit the process. During the monitoring process, the CRO coordinator will check all CRFs and will confirm them to the source documents, and for required cases, the query form will be filled out.

The temperature of the refrigerator which containing the medicines will be checked and recorded by a data logger which will be checked repeatedly by an auditor.

TMF will be checked by CRO coordinator, and it will be rechecked by an auditor. Drug accountability data and information about the proper time for patients' injections will be checked by CRO coordinator and rechecked by sponsor personnel.

After monitoring, problems will be reported by monitor and auditor to the trial centers.

Blinding:

The study will be double-blind. The Subjects and those who conduct the study will be unaware of the state of the patient with regard to the treatment assignments. For this purpose, subjects will be blinded by using a prefilled syringe of Adalimumab, which is quite similar to each other. The injection method, injection syringes, and cartridges are totally the same in both groups. To blind those who conduct the study, the person who delivers or checks the study drug will be different from those who examine the patients. All drugs packages will be identified by unique numbers (manufacture code). Finally, the randomization table will be concealed from research staff by using opaque sealed envelopes.

It should be noted that CRO personnel who enter data into CRF and database and also the sponsor personnel who monitor data entry will be blinded. The study will be double-blind, and situations that might warrant breaking the code are defined in the protocol and include serious adverse events.

Handling of Dropouts or Missing Data:

Since the number of patients who will participate in this clinical trial is limited and small, the investigator can't perform missing imputation analysis and do statistical analysis on those patients who are completed the entire study. However, analyses of the adverse events will be performed on patients who entered the study.

In this study, patients with at least one adverse event will be included in the report. For each adverse event, data will be summarized using frequencies and percentages and then classifies according to the body system. They will be reported in the form of incidence rate. In other words, patients with any number of Adverse Events will be counted only once in this calculation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-75 years at the time of signing the informed consent form.
* Have been diagnosed as having active rheumatoid arthritis (RA) according to The European League Against Rheumatism criteria
* moderately to severely active RA for at least six months
* Patients who have an inadequate response to the treatment with the usual non-biological regimen for at least 12 weeks according to their investigator judgment.
* Ability to comprehend and willingness to sign the Informed Consent Form for this study.

Exclusion Criteria:

* Tuberculosis patient or latent tuberculosis patient (PPD >5mm or abnormal Chest X-ray)
* Have been treated previously with any biological agents including any tumor necrosis factor inhibitors (including ORENCIA® (abatacept), KINERET® (anakinra), REMICADE® (infliximab), ENBREL® (etanercept), CIMZIA® (certolizumab pegol), SIMPONI® (golimumab), or Adalimumab).
* Have a known hypersensitivity to human immunoglobulin proteins or other components of Humira or test- Adalimumab
* Women who are pregnant, breastfeeding or planning to become pregnant during the study
* Have a positive serological test for hepatitis B or hepatitis C or have a known history of infection with human immunodeficiency virus (HIV) of the past three months.
* Physical incapacitation (ACR functional Class IV or wheelchair-/bed-bound)
* Have had a serious infection or have been treated with intravenous antibiotics for an infection within eight weeks or oral antibiotics within two weeks prior to screening
* Have a history of chronic or recurrent infection
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > two times upper limit of normal.
* Hemoglobin <8.5 g/dL.
* Platelets <125,000/µL.
* Leukocyte count <3500/µL.
* Serum Creatinine>2 mg/dl
* Concomitant use of Prednisolone > 10 mg/day and NSAIDs
* Treatment with intravenous, intramuscular, intra-articular and oral corticosteroids within four weeks prior to Day 1 (prednisolone, more than 7.5 mg/daily)
* Ever used RITUXAN® (rituximab), IMURAN® (azathioprine), or PURINETHOL® (mercaptopurine, 6-MP).
* Have any of the following conditions:

  1. History of congestive heart failure.
  2. History of acute myocardial infarction or unstable angina within the previous 12 months prior to Screening.
  3. History of demyelinating disorders (e.g., MS)
  4. History of multiple sclerosis
  5. History of any malignancy within the previous five years prior to Screening.
  6. Any other disease or disorder which, in the opinion of the Investigator, will put the subject at risk if they are enrolled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2016-08-17 (Actual); Study Completion 2017-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmadreza Jamshidi, Professor, Principal Investigator — Rheumatology Research Center, Tehran University of Medical Sciences, Tehran, Iran
Locations (10):
- Iran (10):
  - Alzahra Hospital, Isfahan
  - Besat 4 Clinic, Kerman
  - Ghaem Hospital, Mashhad
  - Razi Hospital, Rasht
  - Imam Ali Clinic, Shahr-e Kord
  - Hafez Hospital, Shiraz
  - Noor Medical Complex, Tabriz
  - Imam Reza Hospital (501 Artesh), Tehran
  - Iran Rheumatism Center, Tehran
  - Loghman Hakim Hospital, Tehran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McInnes IB, Schett G. The pathogenesis of rheumatoid arthritis. N Engl J Med. 2011 Dec 8;365(23):2205-19. doi: 10.1056/NEJMra1004965. No abstract available. PMID 22150039
- [Background] den Broeder A, van de Putte L, Rau R, Schattenkirchner M, Van Riel P, Sander O, Binder C, Fenner H, Bankmann Y, Velagapudi R, Kempeni J, Kupper H. A single dose, placebo controlled study of the fully human anti-tumor necrosis factor-alpha antibody adalimumab (D2E7) in patients with rheumatoid arthritis. J Rheumatol. 2002 Nov;29(11):2288-98. PMID 12415583
- [Background] Singh JA, Furst DE, Bharat A, Curtis JR, Kavanaugh AF, Kremer JM, Moreland LW, O'Dell J, Winthrop KL, Beukelman T, Bridges SL Jr, Chatham WW, Paulus HE, Suarez-Almazor M, Bombardier C, Dougados M, Khanna D, King CM, Leong AL, Matteson EL, Schousboe JT, Moynihan E, Kolba KS, Jain A, Volkmann ER, Agrawal H, Bae S, Mudano AS, Patkar NM, Saag KG. 2012 update of the 2008 American College of Rheumatology recommendations for the use of disease-modifying antirheumatic drugs and biologic agents in the treatment of rheumatoid arthritis. Arthritis Care Res (Hoboken). 2012 May;64(5):625-39. doi: 10.1002/acr.21641. No abstract available. PMID 22473917
- [Background] Keystone EC, Kavanaugh AF, Sharp JT, Tannenbaum H, Hua Y, Teoh LS, Fischkoff SA, Chartash EK. Radiographic, clinical, and functional outcomes of treatment with adalimumab (a human anti-tumor necrosis factor monoclonal antibody) in patients with active rheumatoid arthritis receiving concomitant methotrexate therapy: a randomized, placebo-controlled, 52-week trial. Arthritis Rheum. 2004 May;50(5):1400-11. doi: 10.1002/art.20217. PMID 15146409
- [Background] Furst DE, Schiff MH, Fleischmann RM, Strand V, Birbara CA, Compagnone D, Fischkoff SA, Chartash EK. Adalimumab, a fully human anti tumor necrosis factor-alpha monoclonal antibody, and concomitant standard antirheumatic therapy for the treatment of rheumatoid arthritis: results of STAR (Safety Trial of Adalimumab in Rheumatoid Arthritis). J Rheumatol. 2003 Dec;30(12):2563-71. PMID 14719195
- [Background] Weinblatt ME, Keystone EC, Furst DE, Moreland LW, Weisman MH, Birbara CA, Teoh LA, Fischkoff SA, Chartash EK. Adalimumab, a fully human anti-tumor necrosis factor alpha monoclonal antibody, for the treatment of rheumatoid arthritis in patients taking concomitant methotrexate: the ARMADA trial. Arthritis Rheum. 2003 Jan;48(1):35-45. doi: 10.1002/art.10697. PMID 12528101
- [Background] Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, Katz LM, Lightfoot R Jr, Paulus H, Strand V, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995 Jun;38(6):727-35. doi: 10.1002/art.1780380602. PMID 7779114
- [Background] Scallon B, Cai A, Solowski N, Rosenberg A, Song XY, Shealy D, Wagner C. Binding and functional comparisons of two types of tumor necrosis factor antagonists. J Pharmacol Exp Ther. 2002 May;301(2):418-26. doi: 10.1124/jpet.301.2.418. PMID 11961039
- [Background] Khan MOA, Mohiuddin E, Usmanghani K, Hannan A, Akram M, Shah SA, et al. Clinical evaluation of herbal medicines for the treatment of rheumatoid arthritis. Pak J Nutr. 2011;10(1):51-3.
- [Background] Longo DL, Fauci AS, Kasper DL, Hauser SL, Jameson JL, Loscalzo J. Harrison's principles of internal medicine 18E Vol 2 EB: McGraw Hill Professional; 2012.
- [Background] Alamanos Y, Voulgari PV, Drosos AA. Incidence and prevalence of rheumatoid arthritis, based on the 1987 American College of Rheumatology criteria: a systematic review. Semin Arthritis Rheum. 2006 Dec;36(3):182-8. doi: 10.1016/j.semarthrit.2006.08.006. Epub 2006 Oct 11. PMID 17045630
- [Background] Yood RA, Guidelines ACoRSoRA. Guidelines for the management of rheumatoid arthritis: 2002 update. 2002.
- [Background] Lee WY, Chen HY, Chen KC, Chen CY. Treatment of rheumatoid arthritis with traditional chinese medicine. Biomed Res Int. 2014;2014:528018. doi: 10.1155/2014/528018. Epub 2014 Jun 4. PMID 24991562
- [Background] Weinblatt ME, Schiff M, Valente R, van der Heijde D, Citera G, Zhao C, Maldonado M, Fleischmann R. Head-to-head comparison of subcutaneous abatacept versus adalimumab for rheumatoid arthritis: findings of a phase IIIb, multinational, prospective, randomized study. Arthritis Rheum. 2013 Jan;65(1):28-38. doi: 10.1002/art.37711. PMID 23169319
- [Background] Westhovens R, Kremer JM, Moreland LW, Emery P, Russell AS, Li T, Aranda R, Becker JC, Qi K, Dougados M. Safety and efficacy of the selective costimulation modulator abatacept in patients with rheumatoid arthritis receiving background methotrexate: a 5-year extended phase IIB study. J Rheumatol. 2009 Apr;36(4):736-42. doi: 10.3899/jrheum.080813. Epub 2009 Feb 27. PMID 19273451
- [Background] Navarro Coy NC, Brown S, Bosworth A, Davies CT, Emery P, Everett CC, Fernandez C, Gray JC, Hartley S, Hulme C, Keenan AM, McCabe C, Redmond A, Reynolds C, Scott D, Sharples LD, Pavitt S, Buch MH. The 'Switch' study protocol: a randomised-controlled trial of switching to an alternative tumour-necrosis factor (TNF)-inhibitor drug or abatacept or rituximab in patients with rheumatoid arthritis who have failed an initial TNF-inhibitor drug. BMC Musculoskelet Disord. 2014 Dec 23;15:452. doi: 10.1186/1471-2474-15-452. PMID 25539805
- [Background] Hallikainen A, Vartiainen T. Food control surveys of polychlorinated dibenzo-p-dioxins and dibenzofurans and intake estimates. Food Addit Contam. 1997 May-Jun;14(4):355-66. doi: 10.1080/02652039709374538. PMID 9205564
- [Background] Blumenauer B, Judd M, Cranney A, Burls A, Coyle D, Hochberg M, Tugwell P, Wells G. Etanercept for the treatment of rheumatoid arthritis. Cochrane Database Syst Rev. 2003;(4):CD004525. doi: 10.1002/14651858.CD004525. PMID 14584021
- [Result] Jamshidi A, Gharibdoost F, Vojdanian M, Soroosh SG, Soroush M, Ahmadzadeh A, Nazarinia MA, Mousavi M, Karimzadeh H, Shakibi MR, Rezaieyazdi Z, Sahebari M, Hajiabbasi A, Ebrahimi AA, Mahjourian N, Rashti AM. A phase III, randomized, two-armed, double-blind, parallel, active controlled, and non-inferiority clinical trial to compare efficacy and safety of biosimilar adalimumab (CinnoRA(R)) to the reference product (Humira(R)) in patients with active rheumatoid arthritis. Arthritis Res Ther. 2017 Jul 20;19(1):168. doi: 10.1186/s13075-017-1371-4. PMID 28728599

RESULTS

PARTICIPANT FLOW:
Groups:
- CinnaGen Adalimumab: CinnoRA® (adalimumab Prefilled Syringe produced by CinnaGen Company) 40 mg/0.8 ml Every other week 40 mg Adalimumab will be subcutaneously administered to rheumatic patients during six months. Along with, 15 mg weekly methotrexate, at least 1 mg daily Folic acid and 7.5 mg daily Prednisolone over six months.
  Adalimumab: 40 mg Adalimumab every other week is administered subcutaneously to all the patients.
  Methotrexate: 15 mg Methotrexate is weekly administered to all the patients.
  Folic Acid: At least 1 mg Folic acid is daily administered to all the patients.
  Prednisolone: 7.5 mg Prednisolone is daily administered to all the patients.
- AbbVie Adalimumab: Humira® (adalimumab Prefilled Syringe produced by AbbVie Company) 40 mg/0.8 ml Every other week 40 mg Adalimumab will be subcutaneously administered to rheumatic patients during six months. Along with, 15 mg weekly methotrexate, at least 1 mg daily Folic acid and 7.5 mg daily Prednisolone over six months.
  Adalimumab: 40 mg Adalimumab every other week is administered subcutaneously to all the patients.
  Methotrexate: 15 mg Methotrexate is weekly administered to all the patients.
  Folic Acid: At least 1 mg Folic acid is daily administered to all the patients.
  Prednisolone: 7.5 mg Prednisolone is daily administered to all the patients.
Period: Overall Study
Arm/Group | CinnaGen Adalimumab | AbbVie Adalimumab
Started | 68 | 68
Completed | 64 | 64
Not Completed | 4 | 4
Not completed — Adverse Event | 2 | 3
Not completed — Positive PPD | 1 | 0
Not completed — Poor Compliance | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CinnaGen Adalimumab | AbbVie Adalimumab | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 63 | 122
  >=65 years | 9 | 5 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.29 (12.72) | 47.59 (11.48) | 47.94 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 60 | 118
  Male | 10 | 8 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  Iran | 68 | 68 | 136
Patient assessment of pain [Mean (Standard Deviation); unit: units on a scale] — We used a visual analogue scale (VAS) ranging from 0 (no pain) to 100 (worst possible pain) to assess the "patient assessment of pain".
  units on a scale | 67.21 (23.51) | 70.22 (21.93) | 68.71 (22.70)
Physician's global assessment of disease activity [Mean (Standard Deviation); unit: units on a scale] — We used a visual analogue scale (VAS) ranging from 0 (no disease activity) to 100 (Extremely active disease) to assess the "Physician's global assessment of disease activity".
  units on a scale | 68.97 (17.38) | 70.44 (17.68) | 69.71 (17.48)
Patient global assessment of disease activity [Mean (Standard Deviation); unit: units on a scale] — We used a visual analogue scale (VAS) ranging from 0 (no disease activity) to 100 (Extremely active disease) to assess the "patient global assessment of disease activity".
  units on a scale | 70.15 (20.35) | 70.74 (22.21) | 70.44 (21.23)
Swollen joint count, 28 joints [Mean (Standard Deviation); unit: Swollen joints] | 9.96 (7.39) | 9.46 (6.98) | 9.71 (7.17)
Tender joint count, 28 joints [Mean (Standard Deviation); unit: Tender joints] | 9.46 (8.23) | 9.66 (7.97) | 9.56 (8.08)
Erythrocyte Sedimentation Rate (ESR) [Mean (Standard Deviation); unit: mm/h] | 32.65 (21.24) | 31.12 (24.01) | 31.88 (22.60)
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/L] | 21.40 (25.98) | 18.90 (23.90) | 20.12 (24.87)
DAS28-ESR [Mean (Standard Deviation); unit: units on a scale] — We used the Disease Activity Score-28 for rheumatoid arthritis with erythrocyte sedimentation rate (DAS28-ESR) to assess disease activity in patients with rheumatoid arthritis. This score ranges from 2 to 10, and higher values indicate higher disease activity. DAS28-ESR is calculated with the following formula:
  DAS28-ESR= (0.56*√(Tender Joint Count)+0.28*√(Swollen Joint Count)+0.7*ln(ESR)+0.014*(global health))
  units on a scale | 5.51 (1.24) | 5.47 (1.28) | 5.49 (1.26)
Health Assessment Questionnaire (HAQ) Disability Index [Median (Inter-Quartile Range); unit: units on a scale] — The disability index of Health Assessment Questionnaire (HAQ) is reported which is a self-reported scale to assess the quality of life in rheumatoid arthritis-related studies which includes areas such as dressing/grooming, arising, eating, walking, reach, grip, maintaining hygiene, and daily activities. There are 20 questions in the mentioned 8 sections. In each section, the highest score (between 0 to 3) is considered as the main answer. The final answer is the average of scores relating to all sections. An increased score indicates a worsening of the disability. Population: Because of the missing data in the health assessment questionnaire, row population differs from the overall.
  units on a scale
    number analyzed (Participants) | 65 | 68 | 133
    (all) | 2.25 [1.63 to 3] | 2.38 [1.88 to 3] | 2.38 [1.75 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With DAS28-EULAR Good and Moderate Responses at Week 24
Description: The primary variables are the percentage of patients with DAS28-EULAR Good and Moderate Responses at week 24 compared with Humira. Moderate response is defined as decrement of more than 1.2 in patient's DAS score while patient's DAS score is equal to or more than 3.2 or decrement of 0.6-1.2 while patient's DAS score is equal to or below 5.1. Good response is defined as decrement of more than 1.2 in patient's DAS score while patient's DAS score is below 3.2. We used the Disease Activity Score-28 for rheumatoid arthritis with erythrocyte sedimentation rate (DAS28-ESR) to assess disease activity in patients with rheumatoid arthritis. This score ranges from 2 to 10, and higher values indicate higher disease activity. DAS28-ESR is calculated with the following formula:
  DAS28-ESR= (0.56*√(Tender Joint Count)+0.28*√(Swollen Joint Count)+0.7*ln(ESR)+0.014*(global health))
Time Frame: Week 24
Measure: Number; unit: percentage of participants
Arm/Group | CinnaGen Adalimumab | AbbVie Adalimumab
Number analyzed (Participants) | 64 | 64
percentage of participants | 63 | 63

2. Secondary Outcome: Percentage of Patients Achieving ACR20, ACR50 and ACR70 Response Rates at Week 24
Description: ACR20, ACR50, and ACR70 Response Rates are considered as respectively an Improvement of at Least 20%, 50%, or 70% in American College of Rheumatology (ACR) Score from Baseline at Week 24.
Time Frame: Week 24
Measure: Number; unit: percentage of participants
Arm/Group | CinnaGen Adalimumab | AbbVie Adalimumab
Number analyzed (Participants) | 64 | 64
percentage of participants
  Percentage of Patients achieving ACR20 | 92 | 89
  Percentage of Patients achieving ACR50 | 77 | 75
  Percentage of Patients achieving ACR70 | 47 | 53

3. Secondary Outcome: Health Assessment Questionnaire (HAQ) Disability Index at Week 24.
Description: Quality of life is assessed using the Health Assessment Questionnaire (HAQ). The HAQ is a self-reported scale used in studies of rheumatoid arthritis to assess areas such as dressing/grooming, arising, eating, walking, reach, grip, maintaining hygiene, and daily activities. There are 20 questions in the mentioned 8 sections. In each section, the highest score is considered as the main answer. Scores should be between 0 and 3 and the final answer is the average of scores relating to all sections. An increased score indicates a worsening of the disability. The disability index of Health Assessment Questionnaire (HAQ) at week 24 is reported.
Time Frame: Week 24
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | CinnaGen Adalimumab | AbbVie Adalimumab
Number analyzed (Participants) | 64 | 64
score on a scale | 0.25 [0 to 0.63] | 0.19 [0 to 0.63]

4. Secondary Outcome: The Incidence of Adverse Events
Description: The incidence of adverse events at each visit is recorded based on patients' reports, vital signs, physical examinations, and laboratory tests for systemic safety, including liver function, renal function, complete blood count and clinical chemistries, urinalysis, and hematologic testing.
Time Frame: From the time of first treatment up to the last dose of study treatment; 24 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | CinnaGen Adalimumab | AbbVie Adalimumab
Number analyzed (Participants) | 68 | 68
Participants | 23 | 30

5. Secondary Outcome: Immunogenicity: Number of Participants With Anti-Drug Antibodies (ADA)
Description: Number of Participants with Anti-Drug Antibodies (ADA) at Week 24. The ELISA method was used for immunogenicity assessments of adalimumab.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | CinnaGen Adalimumab | AbbVie Adalimumab
Number analyzed (Participants) | 53 | 55
Participants | 5 | 2

ADVERSE EVENTS:
Arm/Group | CinnaGen Adalimumab | AbbVie Adalimumab
All-Cause Mortality (participants affected / at risk) | 1/68 | 0/68
Serious Adverse Events (participants affected / at risk) | 2/68 | 1/68
Other Adverse Events (participants affected / at risk) | 23/68 | 30/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CinnaGen Adalimumab (N=68) | AbbVie Adalimumab (N=68)
Peritoneal tuberculosis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CinnaGen Adalimumab (N=68) | AbbVie Adalimumab (N=68)
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Injection site reaction (General disorders) | 6 | 12
Respiratory infection (Infections and infestations) | 2 | 7
Sinusitis (Infections and infestations) | 1 | 4
Flu-like symptoms (General disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Headache (Nervous system disorders) | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Urinary tract infection (Infections and infestations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 1
Increased appetite (Metabolism and nutrition disorders) | 2 | 0
Fever (General disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Inflammation localized (General disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Weight increased (Investigations) | 1 | 0
Fatigue (General disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator (PI) may publish results provided a copy of the written publication is received by the sponsor at least 30 days in advance for review and comment. If the parties disagree, PI agrees to meet with the sponsor before submission to resolve any disagreement. It is also agreed that publishing any reports from data is under the condition of the subject's consent. Any reports are highly confidential, and the PI does not have the permission to reveal them without the sponsor's agreement.